CLINICAL TRIAL: NCT05893654
Title: Melphalan Intra-arterial Chemotherapy for Choroidal Melanoma Chemoreduction - a Phase I Clinical Trial
Brief Title: Melphalan Chemoreduction for Ocular Melanoma
Acronym: MELCOM
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital das Clínicas de Ribeirão Preto (Other)
Collaborators: Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48439821100005440
Record Dates: First submitted 2023-05-18; First posted 2023-06-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Uveal Melanoma
Keywords: melanoma; uveal; chemotherapy; chemoreduction; melphalan; ruthenium; brachytherapy
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Melphalan; Brachytherapy; Radiotherapy; Ruthenium-106

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Participants will undergo intra-arterial catheterization of the ophthalmic artery, with administration of 7.5mg of melphalan. After 4±1 weeks, they will receive Ru-106 plaque brachytherapy, which will be performed using a 24-mm notched plaque. Due to tumor thickness and the previous IAC, the target dose to the tumor apex shall be as close as possible to 80 Gy, respecting the safety limits regarding the risk of excessive dosage to the tumor base and scleral melting.
  Interventions: Drug: Melphalan Injection; Radiation: Plaque brachytherapy

INTERVENTIONS:
Drug: Melphalan Injection — 7.5mg of melphalan injected via intra-arterial catheterization of the ophthalmic artery.
  Other Names: Intra-arterial chemotherapy; Chemoreduction
Radiation: Plaque brachytherapy — Brachytherapy will be performed using a 24-mm notched plaque with Ruthenium-106 seeds.
  Other Names: Radiation therapy; Plaque brachytherapy with Ruthenium-106

SUMMARY:
The goal of this clinical trial is to investigate a new approach for treating large uveal melanomas, a type of eye cancer. The study aims to determine the effectiveness of using intra-arterial melphalan, a chemotherapy drug, to reduce tumor thickness, allowing for subsequent radiation therapy using a Ru-106 plaque.

The main questions this trial seeks to answer are:

* Can intra-arterial melphalan effectively reduce the thickness of large uveal melanomas?
* Is the combination of intra-arterial melphalan and brachytherapy a safe and effective treatment option for these tumors?

Participants enrolled in the trial have clinically diagnosed choroidal melanoma with tumor thickness equal to or greater than 8.00 mm. They will undergo a procedure where the chemotherapy drug is injected directly into the blood vessels that supply the tumor. After a few weeks, they will receive the radiation treatment using a small device placed on the eye. Throughout the trial, participants will have different tests to monitor the tumor and their vision, such as ultrasound scans, pictures of the inside of the eye, and a test called electroretinography (ERG) to check the function of the retina. These tests will be done at the start of the trial and at 1, 3, and 6 months later to track the progress of the treatment.

DETAILED DESCRIPTION:
INTRODUCTION Choroidal melanoma is the most common primary intraocular malignancy in adults, thus being the focus of extensive research. The primary treatment goals of this disease consist in controlling local disease, reducing the risk of distant metastases, and avoiding enucleation whenever possible.

Plaque brachytherapy is currently the standard treatment for small and medium-sized uveal melanomas. In clinical practice, ruthenium (Ru-106) or iodine (I-125) are the most commonly employed radioisotopes. Ruthenium is the most utilized radioisotope in Europe and South America due to its availability and good clinical outcomes. It is currently the only available option in Brazil's public health system (SUS). However, its use for large tumors (greater than 10 mm in thickness and/or 22 mm in diameter) is limited by the inability of delivering an adequate therapeutic dose of radiation without causing further damage to the surrounding retinal tissue.

For this reason, researchers in medical physics have been investigating new treatment options in the last decades, including external beam radiotherapy (EBRT), radiosurgery (gamma knife or linear accelerator), and proton beam therapy. Although gamma knife radiosurgery and proton beam therapy are effective treatments with reliable tumor control rates, they are associated with poor visual outcomes, inadequate globe retention, and their use is reportedly limited in public health systems of low- or middle-income countries. EBRT carries potential side effects related to a broader radiation field, with an increased risk for complications in ocular and periocular structures, such as eyelids, sclera, lens, and retina. Finally, enucleation is an effective management for very large tumors, but it is usually a last resource.

Considering the above-mentioned treatment limitations for large choroidal melanomas, our group explored an alternative approach using intra-arterial melphalan for tumor chemoreduction, aiming to reduce thickness and allow subsequent brachytherapy using a Ru-106 plaque.

Intra-arterial chemotherapy (IAC) with melphalan has been used to treat multiple cancers, including liver metastases from uveal and skin melanomas, but it has never been described as a primary tumor treatment. Previous studies have demonstrated a reasonable safety profile of the therapy when used for the treatment of other tumors.

This is a phase I clinical trial that assesses the safety profile of chemoreduction with intra-arterial melphalan, followed by ruthenium brachytherapy, performed in patients that would otherwise need enucleation due to tumor size.

METHODS Patients enrolled in the trial shall have clinically diagnosed choroidal melanoma with tumor thickness equal to or greater than 8.00 mm. IAC with 7.5 mg of melphalan will be performed through selective catheterization of the ophthalmic artery followed by Ru-106 plaque brachytherapy 4±1 weeks after the IAC. All patients will be followed up with baseline and subsequent B-scan ultrasonography, SD-OCT studies, color fundus pictures, infrared photographs, and electroretinograms (ERG).

Baseline and follow-up visits At baseline, patients will undergo a comprehensive ophthalmologic examination including ETDRS best-corrected visual acuity (BCVA), slit lamp biomicroscopy, indirect ophthalmoscopy, spectral-domain optical coherence tomography (SD-OCT), electroretinogram (ERG) performed according to the recommendations of the International Society for Clinical Electrophysiology of Vision (ISCEV) standard,14 and ocular B-scan ultrasound.

OCT examinations will be performed using the Spectralis® HRA+OCT image system (Heidelberg Engineering, Germany). The OCT scan center will be determined at baseline based on patient fixation. In subsequent visits, the automatic follow-up from the Heidelberg machine will be used to scan the same region from the initial visit. Scans over the lesions located close to the posterior pole will also be performed.

Ocular ultrasound will be performed using the Accutome 4sight device in mode B, in the initial consultation, and in 1 month, 3 months, and 6 months after the intervention. The examination will take place with the patient in a seated position, in the most ergonomic and comfortable way as possible, respecting the individual characteristics of the participants.

After the initial assessment, confirmation of the signature of the informed consent, explanation about the procedure, and verbal consent, IAC will be performed in a surgical environment. The intraarterial injection of 7.5 mg of melphalan will be performed only once, in the ophthalmic artery corresponding to the eye affected by choroidal melanoma. Chemotherapy infusion will be performed directly into the ostium of the ophthalmic artery through a microcatheter guided by fluoroscopy via the femoral artery. The drug will be infused in a slow pulsatile manner for 30 minutes to avoid backflow of chemotherapy and arterial occlusion.

After 4±1 weeks, Ru-106 brachytherapy will be performed using a 24-mm notched plaque. Due to tumor thickness and previous IAC, the target dose to the tumor apex should be the closest possible to 80 Gy, respecting the safety limits regarding the risk of excessive dosage to the tumor base and scleral melting.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or higher than 18 years
* Diagnosis of choroidal melanoma with a thickness equal to or higher than 8 mm on ultrasound evaluation
* Comprehension and signature of the informed consent
* Adequate pupil dilation and sufficient cooperation to carry out the complementary exams

Exclusion Criteria:

* Choroidal melanomas with a greatest basal diameter higher than 18mm
* Any clinical condition that impairs fundus documentation or patient follow-up
* Medical or psychological conditions that prevent comprehension and signature of the informed consent
* Pregnancy, breastfeeding, or plans of getting pregnant in the next year
* Past medical history of allergic reactions or hypersensitivity to melphalan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determination of treatment safety through electroretinography (ERG) | 6 months
  Participants will undergo ERG exams at baseline, 1, 3, and 6 months after the first intervention. The researchers will assess the patterns of ERG waves to determine whether there are signs of retinal toxicity.

SECONDARY OUTCOMES:
Reduction of Tumor Size | 6 months
  Measurements of tumor thickness and widest base diameter, in millimeters, as compared to baseline, to be assessed via b-scan ultrasonography.
Best Corrected Visual Acuity (BCVA) | 6 months
  Participants will undergo visual acuity testing at baseline, 1, 3, and 6 months after the first intervention. BCVA will be determined in ETDRS letter changes and the Snellen system.
Signs of intraocular inflammation | 6 months
  Various evaluations including clinical assessment of systemic side effects, B-scan ultrasonography, color fundus pictures, near-infrared photographs, and electroretinography (ERG) will be performed at specific time points: baseline, 1, 3, and 6 months after the first intervention.
Treatment-related adverse events | 6 months
  Participants will be clinically assessed for adverse events immediately after each intervention, as well as 1, 3, and 6 months after the initial intervention. This assessment will be provided by the medical sub-investigators through a thorough anamnesis and clinical examination. Additional investigation, specialty consultations, and laboratory testing may be ordered on an individual basis according to each patient's signs and symptoms.
  We consider an adverse event any untoward medical occurrence or unfavorable sign, symptom, or disease that happens to a participant during the course of the trial, regardless of whether it is related to the interventions being studied. They can encompass a wide range of occurrences, including physical or psychological health problems, abnormal laboratory findings, or worsening of a pre-existing condition.
Globe salvage | 12 months
  Number of enrolled patients that required enucleation or evisceration of the affected eye.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, PhD, Principal Investigator — Professor of Ophthalmology
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting immediately after publication, for an unlimited time.
Access Criteria: Open access.

REFERENCES:
- [Background] Krantz BA, Dave N, Komatsubara KM, Marr BP, Carvajal RD. Uveal melanoma: epidemiology, etiology, and treatment of primary disease. Clin Ophthalmol. 2017 Jan 31;11:279-289. doi: 10.2147/OPTH.S89591. eCollection 2017. PMID 28203054
- [Background] Singh M, Durairaj P, Yeung J. Uveal Melanoma: A Review of the Literature. Oncol Ther. 2018 Jun;6(1):87-104. doi: 10.1007/s40487-018-0056-8. Epub 2018 Feb 6. PMID 32700136
- [Background] American Brachytherapy Society - Ophthalmic Oncology Task Force. Electronic address: paulfinger@eyecancer.com; ABS - OOTF Committee. The American Brachytherapy Society consensus guidelines for plaque brachytherapy of uveal melanoma and retinoblastoma. Brachytherapy. 2014 Jan-Feb;13(1):1-14. doi: 10.1016/j.brachy.2013.11.008. Epub 2013 Dec 24. PMID 24373763
- [Background] Reichstein DA, Brock AL. Radiation therapy for uveal melanoma: a review of treatment methods available in 2021. Curr Opin Ophthalmol. 2021 May 1;32(3):183-190. doi: 10.1097/ICU.0000000000000761. PMID 33770014
- [Background] Parker T, Rigney G, Kallos J, Stefko ST, Kano H, Niranjan A, Green AL, Aziz T, Rath P, Lunsford LD. Gamma knife radiosurgery for uveal melanomas and metastases: a systematic review and meta-analysis. Lancet Oncol. 2020 Nov;21(11):1526-1536. doi: 10.1016/S1470-2045(20)30459-9. PMID 33152286
- [Background] Marinkovic M, Pors LJ, van den Berg V, Peters FP, Schalenbourg A, Zografos L, Pica A, Hrbacek J, Van Duinen SG, Vu THK, Bleeker JC, Rasch CRN, Jager MJ, Luyten GPM, Horeweg N. Clinical Outcomes after International Referral of Uveal Melanoma Patients for Proton Therapy. Cancers (Basel). 2021 Dec 13;13(24):6241. doi: 10.3390/cancers13246241. PMID 34944862
- [Background] Thariat J, Martel A, Matet A, Loria O, Kodjikian L, Nguyen AM, Rosier L, Herault J, Nahon-Esteve S, Mathis T. Non-Cancer Effects following Ionizing Irradiation Involving the Eye and Orbit. Cancers (Basel). 2022 Feb 25;14(5):1194. doi: 10.3390/cancers14051194. PMID 35267502
- [Background] CREECH O Jr, KREMENTZ ET, RYAN RF, WINBLAD JN. Chemotherapy of cancer: regional perfusion utilizing an extracorporeal circuit. Ann Surg. 1958 Oct;148(4):616-32. doi: 10.1097/00000658-195810000-00009. No abstract available. PMID 13583933
- [Background] Hansson J, Lewensohn R, Ringborg U, Nilsson B. Formation and removal of DNA cross-links induced by melphalan and nitrogen mustard in relation to drug-induced cytotoxicity in human melanoma cells. Cancer Res. 1987 May 15;47(10):2631-7. PMID 3567896
- [Background] Minor DR, Allen RE, Alberts D, Peng YM, Tardelli G, Hutchinson J. A clinical and pharmacokinetic study of isolated limb perfusion with heat and melphalan for melanoma. Cancer. 1985 Jun 1;55(11):2638-44. doi: 10.1002/1097-0142(19850601)55:113.0.co;2-e. PMID 3995475
- [Background] Shields CL, Jorge R, Say EA, Magrath G, Alset A, Caywood E, Leahey AM, Jabbour P, Shields JA. Unilateral Retinoblastoma Managed With Intravenous Chemotherapy Versus Intra-Arterial Chemotherapy. Outcomes Based on the International Classification of Retinoblastoma. Asia Pac J Ophthalmol (Phila). 2016 Mar-Apr;5(2):97-103. doi: 10.1097/APO.0000000000000172. PMID 26765038
- [Background] Karydis I, Gangi A, Wheater MJ, Choi J, Wilson I, Thomas K, Pearce N, Takhar A, Gupta S, Hardman D, Sileno S, Stedman B, Zager JS, Ottensmeier C. Percutaneous hepatic perfusion with melphalan in uveal melanoma: A safe and effective treatment modality in an orphan disease. J Surg Oncol. 2018 May;117(6):1170-1178. doi: 10.1002/jso.24956. Epub 2017 Dec 28. PMID 29284076
- [Background] Francis JH, Abramson DH, Gobin YP, Marr BP, Dunkel IJ, Riedel ER, Brodie SE. Electroretinogram monitoring of dose-dependent toxicity after ophthalmic artery chemosurgery in retinoblastoma eyes: six year review. PLoS One. 2014 Jan 20;9(1):e84247. doi: 10.1371/journal.pone.0084247. eCollection 2014. PMID 24465398
- [Background] Robson AG, Frishman LJ, Grigg J, Hamilton R, Jeffrey BG, Kondo M, Li S, McCulloch DL. ISCEV Standard for full-field clinical electroretinography (2022 update). Doc Ophthalmol. 2022 Jun;144(3):165-177. doi: 10.1007/s10633-022-09872-0. Epub 2022 May 5. PMID 35511377